CLINICAL TRIAL: NCT01851252
Title: Pilot Study to Evaluate the Correlation Between ¹³C Methacetin Breath Test (MBT) and HVPG Measurement as a Tool for Identifying Responders to Portal Hypertension Therapy
Brief Title: MBT Versus HVPG in Identifying Responders to Portal Hypertension Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HVPG-BB-EX-513
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Chronic Liver Disease; Cirrhosis; Esophageal Varices; Portal Hypertension; Bleeding
Keywords: Cirrhotics; Esophageal varices; Portal Hypertension
MeSH Terms: conditions — Fibrosis; Esophageal and Gastric Varices; Hypertension, Portal; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methacetin (for BT) before / after Propanolol treatment. (Experimental): The methacetin breath test (MBT) will be performed before and after (within 2 hours) injection of Propanolol (BB) dose and once again after 60 days of oral administration of Propanolol.
  Interventions: Device: Methacetin (with Breath testing device)

INTERVENTIONS:
Device: Methacetin (with Breath testing device) — The methacetin is enriched with carbon 13, a stable non- radioactive isotope, and has been found to be safe in hundreds of studies. The material is very similar to acetominophen. 75 milligrams (mm) of this material pre- dissolved in water are used. This material undergoes rapid metabolism by the liver.

SUMMARY:
The purpose of this study is to determine the effect on the (carbon 13 labelled(13C)-Methacetin Breath Test (MBT) of i.v. propranolol, a non-selective beta blocker (NSBB) following initial administration and after chronic use of each of these agents. The correlation of the MBT with Hepatic Venous Pressure Gradient (HVPG) measurement before and after treatment will be assessed. Additionally, the MBT measurements following 60 days of therapy will be compared to the first MBT measurement and to the second MBT measurement, post HVPG. Each patient's subsequent MBT measurement will be compared to his previous MBT results in order to determine his/her response to therapy.

DETAILED DESCRIPTION:
Variceal bleeding is a life threatening complication of cirrhosis, which still carries a high mortality. Non selective beta-adrenergic blockers are effective at preventing first time variceal bleeding and re-bleeding. The efficacy of these drugs depends on the magnitude of reduction in portal pressure after administration, which varies widely between patients. Studies have shown that a reduction in portal pressure (as measured by HVPG) to 20% from baseline or to values ≤ 12 millimeters of mercury (mmHg) is associated with a low residual risk of bleeding . Patients with such a reduction are considered to be "responders" to beta blocker (BB) therapy. Unfortunately, a significant percentage of patients do not respond to therapy and need to be prescribed to an alternative therapy. The clinical application of this observation is limited since it requires a repeated HVPG measurement,which is not feasible in most cases. A non-invasive breath test that can assess portal pressure in correlation to HVPG and allow efficient management of patients at risk, could be very useful.

ELIGIBILITY:
Inclusion Criteria:

-> 18 years old (M/F)

-Diagnosis of cirrhosis: i. By liver biopsy ii. Or strong suspicion of cirrhosis by accepted criteria for the clinical diagnosis of cirrhosis (e.g. peripheral edema or varices, palpable hard left lobe of the liver, small right lobe span or palpable splenomegaly), and/or radiological evidence of cirrhosis (by abdominal US, CT, or MRI, showing a nodular liver and/or portosystemic collaterals with portal vein patency and/or ascites and/or splenomegaly, and/or colloid shift on a colloid-isotope liver-spleen scan), and/or laboratory variables (platelets <100,000/mm3, albumin< 3.5g/dL, or international normalized ratio (INR)>1.3) iii. Presence of esophageal varices (without previous variceal bleeding episode) or HVPG≥10mmHg 12mmHg from previous testing.

-Has been scheduled for hemodynamic study testing, including response to acute therapy.-

Exclusion Criteria:

* Patients already receiving beta blockers
* Hepatocellular carcinoma
* Portal vein thrombosis
* Contraindications to non-selective beta blocker Propanolol
* Cholestatic liver disease
* Severe heart, pulmonary or renal disease.
* Patient has previous surgical bypass surgery for morbid obesity
* Patient has extensive small bowel resection
* Any major surgery in the past 3 months.
* Patient is a recipient of any organ transplant
* Patient allergic to acetaminophen.
* Patients who are taking hepatotoxic drugs
* Patient, based on the opinion of the investigator, should not be enrolled into this study.
* Patients unable or unwilling to sign informed consent
* Patients that are participating in other clinical trials evaluating experimental treatments or procedures or have participated in a clinical trial in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Correlation between HVPG and MBT and their changes following the i.v. administration of Propranolol | 7 days
  MBT baseline measure will be measured within a week before the anticipated HVPG procedure, but not on the same day. The HVPG will be measured approximately 30 minutes after i.v. propanolol is given and the MBT will be performed approximately one hour later.
The changes between MBT at baseline level and after chronic treatment in Propranolol | 7 days
  MBT baseline measure will be measured within a week before the anticipated HVPG procedure, but not on the same day. The HVPG will be measured approximately 30 minutes after i.v. propanolol is given and the MBT will be performed approximately one hour later.
MBT correlation to clinical events after 2 month of treatment | 67 days
  The MBT will be performed on subjects again after 60 days of oral beta blocker treatment and its results will be compared to previous MBT values.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Ashkenazi, M.D., Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

REFERENCES:
- [Background] Chalasani N, Kahi C, Francois F, Pinto A, Marathe A, Bini EJ, Pandya P, Sitaraman S, Shen J. Improved patient survival after acute variceal bleeding: a multicenter, cohort study. Am J Gastroenterol. 2003 Mar;98(3):653-9. doi: 10.1111/j.1572-0241.2003.07294.x. PMID 12650802
- [Background] Carbonell N, Pauwels A, Serfaty L, Fourdan O, Levy VG, Poupon R. Improved survival after variceal bleeding in patients with cirrhosis over the past two decades. Hepatology. 2004 Sep;40(3):652-9. doi: 10.1002/hep.20339. PMID 15349904
- [Background] Stokkeland K, Brandt L, Ekbom A, Hultcrantz R. Improved prognosis for patients hospitalized with esophageal varices in Sweden 1969-2002. Hepatology. 2006 Mar;43(3):500-5. doi: 10.1002/hep.21089. PMID 16496319
- [Background] de Franchis R. Evolving consensus in portal hypertension. Report of the Baveno IV consensus workshop on methodology of diagnosis and therapy in portal hypertension. J Hepatol. 2005 Jul;43(1):167-76. doi: 10.1016/j.jhep.2005.05.009. No abstract available. PMID 15925423
- [Background] Ripoll C, Groszmann R, Garcia-Tsao G, Grace N, Burroughs A, Planas R, Escorsell A, Garcia-Pagan JC, Makuch R, Patch D, Matloff DS, Bosch J; Portal Hypertension Collaborative Group. Hepatic venous pressure gradient predicts clinical decompensation in patients with compensated cirrhosis. Gastroenterology. 2007 Aug;133(2):481-8. doi: 10.1053/j.gastro.2007.05.024. Epub 2007 May 21. PMID 17681169
- [Background] Abraldes JG, Tarantino I, Turnes J, Garcia-Pagan JC, Rodes J, Bosch J. Hemodynamic response to pharmacological treatment of portal hypertension and long-term prognosis of cirrhosis. Hepatology. 2003 Apr;37(4):902-8. doi: 10.1053/jhep.2003.50133. PMID 12668985
- [Background] Turnes J, Garcia-Pagan JC, Abraldes JG, Hernandez-Guerra M, Dell'Era A, Bosch J. Pharmacological reduction of portal pressure and long-term risk of first variceal bleeding in patients with cirrhosis. Am J Gastroenterol. 2006 Mar;101(3):506-12. doi: 10.1111/j.1572-0241.2006.00453.x. PMID 16542287
- [Background] Groszmann RJ, Bosch J, Grace ND, Conn HO, Garcia-Tsao G, Navasa M, Alberts J, Rodes J, Fischer R, Bermann M, et al. Hemodynamic events in a prospective randomized trial of propranolol versus placebo in the prevention of a first variceal hemorrhage. Gastroenterology. 1990 Nov;99(5):1401-7. doi: 10.1016/0016-5085(90)91168-6. PMID 2210246
- [Background] Feu F, Garcia-Pagan JC, Bosch J, Luca A, Teres J, Escorsell A, Rodes J. Relation between portal pressure response to pharmacotherapy and risk of recurrent variceal haemorrhage in patients with cirrhosis. Lancet. 1995 Oct 21;346(8982):1056-9. doi: 10.1016/s0140-6736(95)91740-3. PMID 7564785
- [Background] Merkel C, Bolognesi M, Sacerdoti D, Bombonato G, Bellini B, Bighin R, Gatta A. The hemodynamic response to medical treatment of portal hypertension as a predictor of clinical effectiveness in the primary prophylaxis of variceal bleeding in cirrhosis. Hepatology. 2000 Nov;32(5):930-4. doi: 10.1053/jhep.2000.19322. PMID 11050041
- [Background] Bureau C, Peron JM, Alric L, Morales J, Sanchez J, Barange K, Payen JL, Vinel JP. "A La Carte" treatment of portal hypertension: Adapting medical therapy to hemodynamic response for the prevention of bleeding. Hepatology. 2002 Dec;36(6):1361-6. doi: 10.1053/jhep.2002.36945. PMID 12447860
- [Background] Bosch J, Groszmann RJ. Measurement of azygos venous blood flow by a continuous thermal dilution technique: an index of blood flow through gastroesophageal collaterals in cirrhosis. Hepatology. 1984 May-Jun;4(3):424-9. doi: 10.1002/hep.1840040312. PMID 6609870
- [Background] Escorsell A, Bordas JM, Castaneda B, Llach J, Garcia-Pagan JC, Rodes J, Bosch J. Predictive value of the variceal pressure response to continued pharmacological therapy in patients with cirrhosis and portal hypertension. Hepatology. 2000 May;31(5):1061-7. doi: 10.1053/he.2000.6779. PMID 10796880
- [Background] Garcia-Tsao G, Grace ND, Groszmann RJ, Conn HO, Bermann MM, Patrick MJ, Morse SS, Alberts JL. Short-term effects of propranolol on portal venous pressure. Hepatology. 1986 Jan-Feb;6(1):101-6. doi: 10.1002/hep.1840060119. PMID 3943775
- [Background] La Mura V, Abraldes JG, Raffa S, Retto O, Berzigotti A, Garcia-Pagan JC, Bosch J. Prognostic value of acute hemodynamic response to i.v. propranolol in patients with cirrhosis and portal hypertension. J Hepatol. 2009 Aug;51(2):279-87. doi: 10.1016/j.jhep.2009.04.015. Epub 2009 May 24. PMID 19501930
- [Background] Valla D, Jiron MI, Poynard T, Braillon A, Lebrec D. Failure of haemodynamic measurements to predict recurrent gastrointestinal bleeding in cirrhotic patients receiving propranolol. J Hepatol. 1987 Oct;5(2):144-8. doi: 10.1016/s0168-8278(87)80565-2. PMID 3500973
- [Background] Merkel C, Bolognesi M, Sacerdoti D, Bombonato G, Cavasin L, Gatta A. Disagreement between acute and chronic haemodynamic effects of nadolol in cirrhosis: a pathophysiological interpretation. Aliment Pharmacol Ther. 2005 Sep 1;22(5):433-9. doi: 10.1111/j.1365-2036.2005.02585.x. PMID 16128681
- [Background] Vorobioff J, Picabea E, Villavicencio R, Puccini V, Rossi O, Bordato J, Audano M. Acute and chronic hemodynamic effects of propranolol in unselected cirrhotic patients. Hepatology. 1987 Jul-Aug;7(4):648-53. doi: 10.1002/hep.1840070406. PMID 3610045
- [Background] Banares R, Moitinho E, Matilla A, Garcia-Pagan JC, Lampreave JL, Piera C, Abraldes JG, De Diego A, Albillos A, Bosch J. Randomized comparison of long-term carvedilol and propranolol administration in the treatment of portal hypertension in cirrhosis. Hepatology. 2002 Dec;36(6):1367-73. doi: 10.1053/jhep.2002.36947. PMID 12447861
- [Background] Braden B, Faust D, Sarrazin U, Zeuzem S, Dietrich CF, Caspary WF, Sarrazin C. 13C-methacetin breath test as liver function test in patients with chronic hepatitis C virus infection. Aliment Pharmacol Ther. 2005 Jan 15;21(2):179-85. doi: 10.1111/j.1365-2036.2005.02317.x. PMID 15679768
- [Background] Festi D, Capodicasa S, Sandri L, Colaiocco-Ferrante L, Staniscia T, Vitacolonna E, Vestito A, Simoni P, Mazzella G, Portincasa P, Roda E, Colecchia A. Measurement of hepatic functional mass by means of 13C-methacetin and 13C-phenylalanine breath tests in chronic liver disease: comparison with Child-Pugh score and serum bile acid levels. World J Gastroenterol. 2005 Jan 7;11(1):142-8. doi: 10.3748/wjg.v11.i1.142. PMID 15609414
- [Background] Goetze O, Selzner N, Fruehauf H, Fried M, Gerlach T, Mullhaupt B. 13C-methacetin breath test as a quantitative liver function test in patients with chronic hepatitis C infection: continuous automatic molecular correlation spectroscopy compared to isotopic ratio mass spectrometry. Aliment Pharmacol Ther. 2007 Jul 15;26(2):305-11. doi: 10.1111/j.1365-2036.2007.03360.x. PMID 17593076
- [Background] de Franchis R. Updating consensus in portal hypertension: report of the Baveno III Consensus Workshop on definitions, methodology and therapeutic strategies in portal hypertension. J Hepatol. 2000 Nov;33(5):846-52. doi: 10.1016/s0168-8278(00)80320-7. No abstract available. PMID 11097497
- [Background] Bosch J, Garcia-Pagan JC, Berzigotti A, Abraldes JG. Measurement of portal pressure and its role in the management of chronic liver disease. Semin Liver Dis. 2006 Nov;26(4):348-62. doi: 10.1055/s-2006-951603. PMID 17051449
- [Background] Groszmann RJ, Wongcharatrawee S. The hepatic venous pressure gradient: anything worth doing should be done right. Hepatology. 2004 Feb;39(2):280-2. doi: 10.1002/hep.20062. No abstract available. PMID 14767976